CLINICAL TRIAL: NCT00626366
Title: Distribution of Topical Nasal Medication Within the Nasal Cavity and Sinuses by Radiographic Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 0498-07-FB
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Sinusitis
Keywords: Nasal Spray; Nasal Drop; Intranasal Medication
MeSH Terms: interventions — Iohexol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal spray (Experimental): This arm of the study will contain subjects who will spray 2-4 sprays of a nasal contrast solution in their nares. Following administration of the spray, the subjects will then have a Xoran mini-CAT scan of their sinuses.
  Interventions: Radiation: Sinus CT Scan; Drug: Omnipaque 240 Contrast Solution
- Nasal drop (Experimental): This arm will contain subjects who will place two drops of a nasal contrast solution in each nose. Following administration of the nasal contrast, the subjects will then have a Xoran miniCAT scan of their sinuses.
  Interventions: Radiation: Sinus CT Scan; Drug: Omnipaque 240 mg I/mL

INTERVENTIONS:
Radiation: Sinus CT Scan — Subjects will undergo a Xoran miniCAT scan of their sinuses
Drug: Omnipaque 240 Contrast Solution — Subjects will spray 2-4 drops of half-strength Omnipaque 240 mgI/mL into each nare. Each spray is approximately 0.1 ml.
  Other Names: contrast enhancement
  Arms: Nasal spray
Drug: Omnipaque 240 mg I/mL — Subjects will place two drops of half-strength Omnipaque 240 mg I/mL intranasally to each nose. Each drop is approximately 1 ml.
  Other Names: contrast enhancement
  Arms: Nasal drop

SUMMARY:
The purpose of this study is to determine the distribution of nasal sprays and nasal drops when used.

DETAILED DESCRIPTION:
The purpose of this study is to determine the distribution of nasal sprays and nasal drops when used. The study hypothesizes that nasal drops will reach the frontonasal region more often than nasal sprays.

ELIGIBILITY:
Inclusion Criteria:

* adult able to perform activities of daily living

Exclusion Criteria:

* signs or symptoms of acute or chronic paranasal sinus disease
* history of sinus surgery
* symptomatic deviated septum
* active seasonal allergies
* allergies to contrast
* history of nasal polyposis
* pregnant or breast feeding women
* neck or back problems that would prevent a subject from kneeling on the floor and crouching over
* currently taking metformin or amiodarone
* students or stff under the direct supervision of the investigators
* cognitive impairment
* terminal illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03-12 (Actual); Primary Completion 2009-01-09 (Actual); Study Completion 2009-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin K O'Brien, MD, Principal Investigator — University of Nebraska; Donald Leopold, MD, Study Chair — University of Nebraska
Locations (1):
- ENT Specialist PC of Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Senocak D, Senocak M, Bozan S. Sinonasal distribution of topically applied particles: computerized tomographic detection and the effects of topical decongestion. Otolaryngol Head Neck Surg. 2005 Dec;133(6):944-8. doi: 10.1016/j.otohns.2005.08.024. PMID 16360518
- [Result] Olson DE, Rasgon BM, Hilsinger RL Jr. Radiographic comparison of three methods for nasal saline irrigation. Laryngoscope. 2002 Aug;112(8 Pt 1):1394-8. doi: 10.1097/00005537-200208000-00013. PMID 12172251
- [Result] Wormald PJ, Cain T, Oates L, Hawke L, Wong I. A comparative study of three methods of nasal irrigation. Laryngoscope. 2004 Dec;114(12):2224-7. doi: 10.1097/01.mlg.0000149463.95950.c5. PMID 15564850
- [Result] Boatsman JE, Calhoun KH, Ryan MW. Relationship between rhinosinusitis symptoms and mucociliary clearance time. Otolaryngol Head Neck Surg. 2006 Mar;134(3):491-3. doi: 10.1016/j.otohns.2005.10.045. PMID 16500451
- [Result] Lund VJ, Black JH, Szabo LZ, Schrewelius C, Akerlund A. Efficacy and tolerability of budesonide aqueous nasal spray in chronic rhinosinusitis patients. Rhinology. 2004 Jun;42(2):57-62. PMID 15224630
- [Result] Aukema AA, Fokkens WJ. Chronic rhinosinusitis: management for optimal outcomes. Treat Respir Med. 2004;3(2):97-105. doi: 10.2165/00151829-200403020-00004. PMID 15182211
- [Result] Cannady SB, Batra PS, Citardi MJ, Lanza DC. Comparison of delivery of topical medications to the paranasal sinuses via "vertex-to-floor" position and atomizer spray after FESS. Otolaryngol Head Neck Surg. 2005 Nov;133(5):735-40. doi: 10.1016/j.otohns.2005.07.039. PMID 16274802

RESULTS

PARTICIPANT FLOW:
Groups:
- Nasal Drops: This arm will contain subjects who will place two drops of a nasal contrast solution in each nose. Following administration of the nasal contrast, the subjects will then have a Xoran miniCAT scan of their sinuses.
  Sinus CT Scan: Subjects will undergo a Xoran miniCAT scan of their sinuses
  Omnipaque 240 mg I/mL: Subjects will place two drops of half-strength Omnipaque 240 mg I/mL intranasally to each nose. Each drop is approximately 1 ml.
Period: Overall Study
Arm/Group | Nasal Spray | Nasal Drops
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Spray | Nasal Drops | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.6 [19 to 50] | 28.6 [19 to 50] | 28.6 [19 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: To Measure the Distribution of Nasal Sprays and Drops.
Description: CT scan scored for distribution contrast delivered by nasal spray or drops within subsets in the nasal cavity. The sinonasal cavity was divided into twenty-one subsites on each side of the nasal cavity. The interpreters scored for the presence (1) or absence (0) of contrast from the nasal spray or nasal drops within each subsite. Left and right sides were interpreted separately for a possible total score of 0-42 for each CT scan.
Time Frame: 2 months
Population: Each participant's CT scan will be scored for left and right sides for a total of 18 sinonasal cavities
Measure: Number; unit: nasal cavities (right and left sides)
Units Other Than Participants: nasal cavities (right and left sides)
Arm/Group | Nasal Spray | Nasal Drops
Number analyzed (Participants) | 9 | 9
Number analyzed (nasal cavities (right and left sides)) | 18 | 18
nasal cavities (right and left sides)
  Nasal vestibule | 18 | 17
  Inferior upper nasal vault | 16 | 17
  Superior upper nasal vault | 0 | 6
  Anterior floor of nose | 12 | 4
  Anterior inferior meatus | 16 | 0
  Anterior inferior nasal cavity | 15 | 6
  Posterior floor of nose | 9 | 0
  Posterior inferior meatus | 9 | 1
  Posterior inferior nasal cavity | 3 | 1
  Anterior middle nasal cavity | 3 | 5
  Anterior olfactory cleft | 1 | 4
  Posterior middle nasal cavity | 2 | 4
  Posterior olfactory cleft | 1 | 4
  Anterior middle meatus | 4 | 2
  Anterior ethmoid | 2 | 1
  Osteomeatal complex | 2 | 1
  Posterior middle meatus | 2 | 1
  Posterior ethmoid | 1 | 2
  Frontal recess | 0 | 2
  Sphenoethmoid recess | 2 | 4
  Nasopharynx | 8 | 2

ADVERSE EVENTS:
Arm/Group | Nasal Spray | Nasal Drop
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes